CLINICAL TRIAL: NCT01318512
Title: The Dosage of MIRCERA in the Treatment of Renal Anaemia in Patients With Chronic Renal Disease Who do Not Undergo Haemodialysis in Clinical Practice
Brief Title: An Observational Study of Mircera (Methoxy Polyethylene Glycol-epoetin Beta) in Patients With Chronic Kidney Disease Not On Dialysis
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25317
Record Dates: First submitted 2011-03-17; First posted 2011-03-18 (Estimated); Results first posted 2015-12-03 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-05

CONDITIONS: Kidney Disease, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Chronic Kidney Disease: Participants with CKD, not undergoing haemodialysis in clinical practice setting and started treatment with methoxy polyethylene glycol-epoetin beta (MIRCERA) subcutaneously (SC) as per summary of product characteristics (SPC) due to decreased levels of haemoglobin.

SUMMARY:
This observational, prospective, multicenter study will describe the mean dose of Mircera (methoxy polyethylene glycol-epoetin beta) and the hemoglobin levels in patients with chronic kidney disease. Patients are not on dialysis and are naive to, or have received erythropoiesis stimulating agent treatment. Data will be collected for 10 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients, >/=18 years of age
* Presence of chronic kidney disease (Stage 3-4)

Exclusion Criteria:

* Participation in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic kidney disease receiving Mircera treatment
Sampling Method: Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2010-07-31 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2013-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Nemocnice Novy Jicin; Dialyzacni Stredisko, Nový Jičín, Czechia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study included Titration Period (4 months) and Maintenance Period (6 Months).
Groups:
- Chronic Kidney Disease (CKD): Participants with CKD, not undergoing hemodialysis in clinical practice setting and started treatment with methoxy polyethylene glycol-epoetin beta (MIRCERA) subcutaneously (SC) as per summary of product characteristics (SPC) due to decreased levels of hemoglobin.
Period: Titration Period (4 Months)
Arm/Group | Chronic Kidney Disease (CKD)
Started | 340
Completed | 340
Not Completed | 0
Period: Maintenance Period (6 Months)
Arm/Group | Chronic Kidney Disease (CKD)
Started | 340
Completed | 329
Not Completed | 11
Not completed — Death | 2
Not completed — Protocol Violation | 9

BASELINE CHARACTERISTICS:
Population: All enrolled participants were included.
Arm/Group | Chronic Kidney Disease (CKD)
Number analyzed (Participants) | 340
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 172
  Male | 168

OUTCOME MEASURES:

1. Primary Outcome: Average Dose of MIRCERA at Entry Level
Description: The average dose of MIRCERA, measured in micrograms (µg) at entry level was reported.
Time Frame: Baseline
Population: All participants who received at least one dose of MIRCERA during the titration period.
Measure: Mean (Standard Deviation); unit: microgram (µg)
Groups:
- Chronic Kidney Disease (CKD): Participants with CKD, not undergoing hemodialysis in clinical practice setting and started treatment with MIRCERA subcutaneously due to decreased levels of hemoglobin.
Arm/Group | Chronic Kidney Disease (CKD)
Number analyzed (Participants) | 340
microgram (µg) | 94 (49)

2. Secondary Outcome: The Mean Hemoglobin (Hb) Level During Titration Period
Description: The hemoglobin level was measured in grams per liter (g/L) at entry level and after each month of treatment with MIRCERA. The study did not distinguish between erythropoiesis stimulating agent naive and erythropoiesis stimulating agent treated participants, and collected the overall data (Hb level) before/after administration of MIRCERA.
Time Frame: Baseline, Month 1, 2, 3, 4
Population: All participants who received at least one dose of MIRCERA during titration period.
Measure: Mean (Standard Deviation); unit: g/L
Groups:
- Chronic Kidney Disease (CKD): Participants with CKD, not undergoing haemodialysis in clinical practice setting and started treatment with MIRCERA subcutaneously due to decreased levels of haemoglobin.
Arm/Group | Chronic Kidney Disease (CKD)
Number analyzed (Participants) | 340
g/L
  Baseline | 93.9 (11.7)
  Month 1 | 98.4 (12.4)
  Month 2 | 103.4 (12.7)
  Month 3 | 106.3 (12.0)
  Month 4 | 108.4 (12.4)

3. Secondary Outcome: The Mean Hemoglobin (Hb) Level During Maintenance Period
Description: The hemoglobin level was measured in grams per liter (g/L) after each month of treatment with MIRCERA. The study did not distinguish between erythropoiesis stimulating agent naive and erythropoiesis stimulating agent treated participants, and collected the overall data (Hb level) before/after administration of MIRCERA
Time Frame: Month 5, 6, 7, 8, 9, 10
Population: All participants who received at least one dose of MIRCERA during maintenance period.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Chronic Kidney Disease (CKD)
Number analyzed (Participants) | 340
g/L
  Month 5 | 109.3 (11.6)
  Month 6 | 110.3 (10.3)
  Month 7 | 111.2 (9.8)
  Month 8 | 112.1 (10.3)
  Month 9 | 112.5 (10.9)
  Month 10 | 113.8 (10.9)

4. Primary Outcome: Average Dose of MIRCERA During Titration Period Month 1
Description: The average dose of MIRCERA, measured in microgram (µg) at each month interval during the titration period was reported.
Time Frame: Month 1
Population: All participants who received at least one dose of MIRCERA during titration period.
Measure: Mean (Standard Deviation); unit: microgram (µg)
Arm/Group | Chronic Kidney Disease (CKD)
Number analyzed (Participants) | 340
microgram (µg) | 101.3 (54)

5. Primary Outcome: Average Dose of MIRCERA During Titration Period Month 2
Description: The average dose of MIRCERA, measured in micrograms (µg) at each month interval during the titration period was reported.
Time Frame: Month 2
Population: All participants who received at least one dose of MIRCERA during titration period.
Measure: Mean (Standard Deviation); unit: microgram (µg)
Arm/Group | Chronic Kidney Disease (CKD)
Number analyzed (Participants) | 340
microgram (µg) | 102.4 (54.3)

6. Primary Outcome: Average Dose of MIRCERA During Titration Period Month 3
Description: as for outcome 5
Time Frame: Month 3
Population: All participants who received at least one dose of MIRCERA during titration period.
Measure: Mean (Standard Deviation); unit: microgram (µg)
Arm/Group | Chronic Kidney Disease (CKD)
Number analyzed (Participants) | 340
microgram (µg) | 106.1 (56.2)

7. Primary Outcome: Average Dose of MIRCERA During Titration Period Month 4
Description: as for outcome 5
Time Frame: Month 4
Population: All participants who received at least one dose of MIRCERA during titration period.
Measure: Mean (Standard Deviation); unit: microgram (µg)
Arm/Group | Chronic Kidney Disease (CKD)
Number analyzed (Participants) | 340
microgram (µg) | 107.5 (59.8)

8. Primary Outcome: Average Dose of MIRCERA During Maintenance Period Month 1
Description: The average dose of MIRCERA, measured in micrograms (µg) at each month interval during the maintenance period was reported.
Time Frame: Month 5 (Maintenance Period Month 1)
Population: All participants who received at least one dose of MIRCERA during the maintenance period.
Measure: Mean (Standard Deviation); unit: microgram (µg)
Arm/Group | Chronic Kidney Disease (CKD)
Number analyzed (Participants) | 340
microgram (µg) | 105 (61)

9. Primary Outcome: Average Dose of MIRCERA During Maintenance Period Month 2
Description: as for outcome 8
Time Frame: Month 6 (Maintenance Period Month 2)
Population: All participants who received at least one dose of MIRCERA during the maintenance period.
Measure: Mean (Standard Deviation); unit: microgram (µg)
Arm/Group | Chronic Kidney Disease (CKD)
Number analyzed (Participants) | 340
microgram (µg) | 106 (61.7)

10. Primary Outcome: Average Dose of MIRCERA During Maintenance Period Month 3
Description: as for outcome 8
Time Frame: Month 7 (Maintenance Period Month 3)
Population: All participants who received at least one dose of MIRCERA during the maintenance period.
Measure: Mean (Standard Deviation); unit: microgram (µg)
Arm/Group | Chronic Kidney Disease (CKD)
Number analyzed (Participants) | 340
microgram (µg) | 107 (63.6)

11. Primary Outcome: Average Dose of MIRCERA During Maintenance Period Month 4
Description: as for outcome 8
Time Frame: Month 8 (Maintenance Period Month 4)
Population: All participants who received at least one dose of MIRCERA during the maintenance period.
Measure: Mean (Standard Deviation); unit: microgram (µg)
Arm/Group | Chronic Kidney Disease (CKD)
Number analyzed (Participants) | 340
microgram (µg) | 109 (66.5)

12. Primary Outcome: Average Dose of MIRCERA During Maintenance Period Month 5
Description: as for outcome 8
Time Frame: Month 9 (Maintenance Period Month 5)
Population: All participants who received at least one dose of MIRCERA during the maintenance period.
Measure: Mean (Standard Deviation); unit: microgram (µg)
Arm/Group | Chronic Kidney Disease (CKD)
Number analyzed (Participants) | 340
microgram (µg) | 112 (66.2)

13. Primary Outcome: Average Dose of MIRCERA During Maintenance Period Month 6
Description: as for outcome 8
Time Frame: Month 10 (Maintenance Period Month 6)
Population: All participants who received at least one dose of MIRCERA during the maintenance period.
Measure: Mean (Standard Deviation); unit: microgram (µg)
Arm/Group | Chronic Kidney Disease (CKD)
Number analyzed (Participants) | 340
microgram (µg) | 114 (65.9)

ADVERSE EVENTS:
Time Frame: 3.5 years
Arm/Group | Chronic Kidney Disease (CKD)
Serious Adverse Events (participants affected / at risk) | 5/340
Other Adverse Events (participants affected / at risk) | 2/340
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chronic Kidney Disease (CKD) (N=340)
Cardiac failure left (Cardiac disorders) | 1
Sepsis (Infections and infestations) | 1
Endocarditis infective (Infections and infestations) | 1
Peripheral arterial disease (Vascular disorders) | 1
Post surgical haemorrhage (Injury, poisoning and procedural complications) | 1
Surgery (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chronic Kidney Disease (CKD) (N=340)
Headache (Nervous system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.